CLINICAL TRIAL: NCT06298708
Title: Comparison of Immunogenicity and Safety of Inactivated and Live-attenuated Hepatitis A Virus Vaccine Among Thai Healthy Children and Adolescents: A Randomized, Active-controlled, Open-label, Non-inferiority Trial
Brief Title: Immunogenicity and Safety of Inactivated and Live-attenuated HAV Vaccine Among Thai Healthy Children and Adolescents
Acronym: HAV-RCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Collaborators: Faculty of Medicine, Chiang Mai University (Unknown)
Responsible Party: Principal Investigator, Tavitiya Sudjaritruk, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PED-2566-0634
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: HAV; Hepatitis A; Hep A; Vaccine-Preventable Diseases
Keywords: HAV vaccine; immunogenicity; safety; randomized controlled trial
MeSH Terms: conditions — Hepatitis A; Vaccine-Preventable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-HAV (Experimental): Live-attenuated hepatitis A vaccine.
  Interventions: Biological: Mevac-A vaccine
- I-HAV (Active Comparator): Inactivated hepatitis A vaccine.
  Interventions: Biological: Havrix 720 Junior

INTERVENTIONS:
Biological: Mevac-A vaccine — Mevac-A: A freeze-dried live-attenuated hepatitis A vaccine.
  Dose and administration: a freeze-dried live-attenuated vaccine, subcutaneous injection of 0.5 ml will be administered for 1 time.
  Arms: L-HAV
Biological: Havrix 720 Junior — Havrix 720 Junior: An inactivated hepatitis A vaccine, 720 ELISA units per 0.5 ml of formaldehyde-inactivated hepatitis A virus (HM175 hepatitis A virus strain).
  Dose and administration: a pre-filled syringe, intramuscular injection of 0.5 ml will be administered for 2 times with 6-month interval.
  Arms: I-HAV

SUMMARY:
Hepatitis A virus (HAV) vaccine is an effective strategy to prevent natural HAV infection. In Thailand, there are 2 types of HAV vaccine available, including inactivated HAV vaccine and live-attenuated HAV vaccine. This study aims to compare the immunogenicity and safety of inactivated and lived-attenuated HAV vaccine among Thai healthy children and adolescents age 18 months to 18 years.

DETAILED DESCRIPTION:
Hepatitis A virus (HAV) infection is one of the common cause of viral hepatitis in children and adolescents in developing countries, including Thailand. This virus is easily transmitted through ingestion of contaminated food and water or through direct contact with an infectious person. Generally, HAV causes acute hepatitis, ranging mild illness to severe fulminant hepatitis (acute liver failure), but does not cause chronic liver disease. HAV vaccine is an effective strategy to prevent natural HAV infection as well as serious consequences of the illness.

Currently, there are 2 types of HAV vaccine available in Thailand, including (1) inactivated vaccine (I-HAV) which is recommended for 2 doses, 6 months apart and is approved for children age 1 year and above; and (2) live-attenuated vaccine (L-HAV) which is recommended for 1 dose and is approved for children age 18 months and above. However, these vaccines have not included in the Thailand Expanded Programme on Immunization (EPI) yet. Thus, vaccination coverage rate is suboptimal in the country. Moreover, the information regarding immunogenicity and safety of both vaccines is limited.

This is a randomized, active-controlled, open-label, non-inferiority trial which aims to compare the immunogenicity and safety of a marketed inactivated (I-HAV) and a live-attenuated HAV vaccine (L-HAV) among Thai healthy children and adolescents age 18 months to 18 years. This study will provide important information about the immunogenicity and safety profiles of both vaccines in Thai healthy youth as well as demonstrate the associated factors of HAV vaccine-elicited immunity in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 months and 18 years
* Has healthy status
* Has no history of hepatitis A infection or previous hepatitis A disease
* Has never received hepatitis A vaccine (from vaccine booklet or parental history)
* Participants and/or caregivers gives written inform consent/assent form

Exclusion Criteria:

* Has acute illness within 4 weeks before enrollment
* Has fever with jaundice within 4 weeks before enrollment
* Has underlying disease of thrombocytopenia, coagulopathy, hemophilia A or B, neurologic disease, immunocompromised condition, chronic liver disease, chronic hepatitis B or C infection
* Has received immunosuppressive agents or immunomodulatory agents, corticosteroid >2 mg/kg/day or 20 mg/day within 6 months before enrollment
* Has received blood or blood component, or intravenous immunoglobulin within 6 months before enrollment
* Has received any lived-attenuated vaccine within 30 days before enrollment
* Has history of severe allergy to vaccine or vaccine component, including aluminum hydroxide, 2-phenoxyethanol, neomycin, formaldehyde, gentamicin sulfate, or has history of anaphylaxis or severe allergic reactions following vaccination
* Women planning for pregnancy, pregnant women or lactating women
* Women in childbearing age who cannot use contraceptive methods during study participation
* Is concurrently involved in other clinical trials in which receiving an investigational vaccine or study drug as part of study participation
* Have any condition that, in the opinion of the site investigator, would compromise the subject's ability to participate in the study

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2024-04-27 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Anti-HAV immunoglobulin G (IgG) seroconversion rate | L-HAV group: 4 weeks after the first vaccination. I-HAV group: 4 weeks after the second vaccination
  Anti-HAV IgG seroconversion rate (anti-HAV IgG >= 1.0 S/CO) after the first vaccination for L-HAV group and after the second vaccination for I-HAV group, among participants with anti-HAV IgG <1.0 S/CO at baseline.

SECONDARY OUTCOMES:
Geometric mean concentration (GMC) of anti-HAV IgG level | Baseline (before the first vaccination), 4 weeks after the first vaccination, and 4 weeks after the second vaccination (for I-HAV group only).
  Geometric mean concentration (GMC) of anti-HAV IgG level before the first vaccination, 4 weeks after the first vaccination, and 4 weeks after the second vaccination (for I-HAV group only).

CONTACTS AND LOCATIONS:
Overall Officials: Tavitiya Sudjaritruk, MD, PhD, Study Chair — Department of Pediatrics, Faculty of Medicine, Chiang Mai University; Natchaya Kunanitthaworn, MD, Principal Investigator — Department of Pediatrics, Faculty of Medicine, Chiang Mai University
Locations (1):
- Department of Pediatrics, Faculty of Medicine, Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available for this study.

REFERENCES:
- [Background] Kunanitthaworn N, Mueangmo O, Saheng J, Wongjak W, Lertsiriladakul T, Chaito T, Nantarat P, Sudjaritruk T. Seroprevalence of hepatitis A virus antibodies among children and adolescents living in Northern Thailand: an implication for hepatitis A immunization. Sci Rep. 2023 Oct 13;13(1):17432. doi: 10.1038/s41598-023-44643-0. PMID 37833325
- [Background] Ma F, Yang J, Kang G, Sun Q, Lu P, Zhao Y, Wang Z, Luo J, Wang Z. Comparison of the safety and immunogenicity of live attenuated and inactivated hepatitis A vaccine in healthy Chinese children aged 18 months to 16 years: results from a randomized, parallel controlled, phase IV study. Clin Microbiol Infect. 2016 Sep;22(9):811.e9-811.e15. doi: 10.1016/j.cmi.2016.06.004. Epub 2016 Jun 23. PMID 27345175
- [Background] Liu XE, Wushouer F, Gou A, Kuerban M, Li X, Sun Y, Zhang J, Liu Y, Li J, Zhuang H. Comparison of immunogenicity between inactivated and live attenuated hepatitis A vaccines: a single-blind, randomized, parallel-group clinical trial among children in Xinjiang Uighur Autonomous Region, China. Hum Vaccin Immunother. 2013 Jul;9(7):1460-5. doi: 10.4161/hv.24366. Epub 2013 Apr 9. PMID 23571173